CLINICAL TRIAL: NCT00207506
Title: HoMBReS: A Lay Health Advisor Approach to Sexually Transmitted Disease Prevention
Brief Title: Lay Health Advisors for Sexually Transmitted Disease Prevention
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-4337; U36/CCU300860
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Syphilis; Gonorrhea; Chlamydia Infections; HIV Infections
Keywords: Latino; Lay Health; Access; Prevention; HIV Seronegativity; HIV
MeSH Terms: conditions — Syphilis; Gonorrhea; Chlamydia Infections; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: HoMBReS: A lay health advisor approach to STD prevention

SUMMARY:
Non-professional community leaders may be at a great advantage in reaching otherwise hard to reach populations for the purpose of advising on sexually transmitted disease (STD) prevention (lay health advisors), health care access, and model health behavior. Latino migrant farm workers are at increased risk for STD and might benefit from such lay health advisors. The study will examine whether this strategy is a useful one for STD prevention in Latino migrant farm workers in rural and small town areas of North Carolina.

DETAILED DESCRIPTION:
This is a demonstration project which includes the development, implementation, and evaluation of HoMBReS: Hombres Manteniendo Bienestar y Relaciones Saludables (Men Maintaining Wellness and Healthy Relationships). Applying a community-based participatory research (CBPR) approach, this 3-year study uses a quasi-experimental delayed-intervention comparison group design to assess the feasibility of implementing and the potential efficacy of an adult soccer league-based lay health advisor intervention. The intervention is designed to: reduce sexual risk behaviors among Latino seasonal farmworkers; enhance access to sexually transmitted disease/HIV healthcare services; and develop effective data collection methods among Latino men.

ELIGIBILITY:
Inclusion Criteria:

LHA (lay health advisor) and participants:

* To be eligible for participation in this study as a lay health advisor (LHA), an LHA must:

  1. self-identify as Latino or Hispanic;
  2. work as a migrant or seasonal farmworker;
  3. be a member of the Liga Hispana de Fútbol de NC;
  4. be 18 years of age;
  5. be literate in Spanish; and
  6. provide informed consent.

Exclusion Criteria:

* Based on the characteristics of the league population, the researchers anticipate that few potential LHAs or participants will be excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2004-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Reduced STD morbidity
Reduced risk behavior

SECONDARY OUTCOMES:
Improved access to services

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rhodes, PhD, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States